CLINICAL TRIAL: NCT03654495
Title: Neuroplasticity Associated With Anterior Cruciate Ligament Injury: A Single Centre, Cross-sectional Observational & Usual-care-controlled Pilot-RCT Assessing a Motor Learning Based Therapy Intervention
Brief Title: Neuroplasticity Associated With Anterior Cruciate Ligament Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Eling DeBruin, Professor, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC-Nr. 2017-01925; ACL-ETH-2017 (Registry Identifier: BASEC)
Record Dates: First submitted 2018-07-17; First posted 2018-08-31 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: This trial is a two-arm, parallel-group, randomized-controlled pilot trial with a cross-sectional comparison at baseline.
Masking Description: The aim is to focus on recruitment, attrition and adherence to the rehabilitation intervention. This trial is composed of a comparative cross-sectional part and a randomized conventional rehabilitation-controlled trial part with 1:1 allocation ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame Training (Experimental): Routine (standard) therapy given based on conventional current-best-evidence Rehabilitation. In addition training on Medical Device (MD): Dividat Senso, DIV-SENSO-H, Dividat GmbH, Software development: ISO 62304:2016; designed to train different aspects of executive functions (EFs; divided attention, working memory, inhibition, and shifting) and physical functions through Virtual Reality video game training.
  Interventions: Other: Exergame training; Other: Usual Care Training
- Usual Care Training (Active Comparator): Routine (standard) therapy given based on conventional current-best-evidence Rehabilitation.
  Interventions: Other: Usual Care Training

INTERVENTIONS:
Other: Exergame training — Training on Medical Device (MD): Dividat Senso, DIV-SENSO-H, Dividat GmbH, Software development: ISO 62304:2016; designed to train aspects of executive functions (EFs; divided attention, working memory, inhibition, and shifting) and physical functions through Virtual Reality video game training.
  FITT training principles are implemented; Frequency: three times per week, Intensity: individually adapted VG (allowing training progression), Type: combination of cognitive and motor training, and Time: 20 min training sessions. Training lasts 6 weeks (18 training sessions). Participants train 20 min, three times per week. Training includes one session of each VG (4 min) in a pre-defined order and short breaks (~1 min) for game change.
  Arms: Exergame Training
Other: Usual Care Training — Routine (standard) therapy given based on conventional current-best-evidence Rehabilitation. Preoperative Phase: Diminish inflammation, swelling, and pain; Restore normal range of motion (especially knee extension); Restore voluntary muscle activation Immediate Postoperative Phase (Day 1-7): Restore full passive knee extension; Diminish joint swelling and pain; Restore independent ambulation Early Rehabilitation Phase (Week 2-4): Maintain full passive knee extension; Gradually increase knee flexion; Muscle training Controlled Ambulation Phase (Week 4-10): Restore full knee ROM; Improve lower extremity strength; Enhance proprioception, balance, and neuromuscular control Advanced Activity Phase (Week 10-16): Normalize lower extremity strength; Enhance muscular power and endurance; Improve neuromuscular control; Perform selected sport-specific drills.

SUMMARY:
Activation of the brain for knee movement changes after anterior cruciate ligament (ACL) reconstruction. The brain activation profile after ACL reconstruction indicates a shift to a visual-motor control strategy, as opposed to a sensory-motor control strategy to control the knee movement. Recent research suggests that ACL reconstruction rehabilitation protocols should also consider neurocognition and its role in exercise, neuromuscular control, and injury risk to improve the effectiveness of the intervention.

However, there is currently no evidence of the feasibility of neurocognitive exercise in a primary rehabilitation program that aims to restore movement function after ACL damage.

The purpose of this study is to assess whether conventional ACL injury training with additional cognitive training based on virtual reality is as effective as the sole conventional ACL injury training in participants with ACL injuries.

DETAILED DESCRIPTION:
Whereas three percent of amateur athletes injure their anterior cruciate ligament (ACL) each year, this percentage can be as high as 15% in elite athletes. Because the ACL contains mechanoreceptors it directly influences the neuromuscular control of the knee. ACL deficiency leads to partial deafferentiation which, in turn, alters spinal and supraspinal motor control.

Return to sports following ACL injuries is mostly decided based on time since surgery; however, this decision process produces unsuccessful outcomes; e.g. high re-injury rates or athletes not being able to return to their pre-injury sport levels. The rate of return to preinjury play levels for non-professional pivoting athletes for example is 65%. A recent evidence-based clinical update revealed that it is currently unclear whether there is a benefit of supervised physical therapy rehabilitation compared to home-based rehabilitation or no rehabilitation at all, and comparisons between 19-week with 32-week rehabilitation programmes show no differences in terms of laxity, range of motion, knee function, or measures of leg muscle strength. Evidence-based guidelines suggest practitioners should generally follow a moderate recommendation, which means that the benefits of treatment exceed the potential harm; however, the quality/applicability of the supporting evidence is not as strong. Many rehabilitation programs currently target biomechanical factors; e.g. muscle strength, balance and plyometric function, and consider to a rather lesser extend cognitive or neurological components.

Brain activation for knee flexion/extension motion alters following ACL reconstruction. The brain activation profile following ACL reconstruction may indicate a shift toward a visual-motor strategy as opposed to a sensory-motor strategy to engage in knee movement. This recent research evidence suggests that rehabilitation protocols for ACL reconstruction should additionally be considering neurocognition and its role in movement, neuromuscular control, and injury risk to help improve intervention effectiveness.

However, there is a lack of evidence concerning the feasibility of implementing neurocognitive exercise interventions in a primary rehabilitation program aimed at restoring function following ACL injury. New treatments usually have to go through a series of phases to test whether they are safe and effective before larger scale studies and application in clinical practice are to be considered. The aim of this pilot study was to perform a phase II trial according the model for complex interventions advocated by the British Medical Research Council to test the feasibility and effects of a conventional ACL injury rehabilitation program with added neurocognitive training in a group of ACL injured individuals. This study aims to: (1) compare ACL injured individuals with non-injured individuals, (2) develop an exercise intervention based on research literature theory and to deliver it to ACL injured individuals, (3) evaluate the feasibility of the intervention and the ability to recruit and retain ACL injured individuals, and (4) assess whether the treatment has some effect on neural drive and physical performance.

ELIGIBILITY:
The inclusion criteria for the cross-sectional study part are:

* 18- to 55-year-old subjects
* healthy or in the subacute phase (from 7 to 21 days) or in the chronic phase (≥ one year) after unilateral surgical reconstruction of complete ACL rupture, confirmed by MRI in the medical record and by the surgical procedure.

The exclusion criteria for the cross-sectional study part are:

* not healthy
* bilaterally previous diagnoses in the medical record, such as neuropathic pain in the lower limb, lumbosacral radiculopathy, saphenous nerve entrapment, meralgia paresthetica, fractures, rheumatoid or systemic conditions, other surgeries, post-surgery complications (i.e., thrombosis or osteomyelitis), belonephobia, legs length difference in the lower limb (>0.5 cm) [https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5413255/].

The inclusion criteria for the longitudinal study part are:

• 18- to 55-year-old subjects, in the subacute phase (from 7 to 21 days) after unilateral surgical reconstruction of complete ACL rupture, confirmed by MRI in the medical record and by the surgical procedure.

The exclusion criteria for the longitudinal study part are:

• bilaterally previous diagnoses in the medical record, such as neuropathic pain in the lower limb, lumbosacral radiculopathy, saphenous nerve entrapment, meralgia paresthetica, fractures, rheumatoid or systemic conditions, other surgeries, post-surgery complications (i.e., thrombosis or osteomyelitis), belonephobia, legs length difference in the lower limb (>0.5 cm) [https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5413255/].

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Attrition; number of participants lost at follow-up | six weeks
  For recruitment, data for the total sampling frame (both those approached and not approached) for inclusion in the trial is taken to assess generalizability to ACL individuals. This will be assessed at the end of the 6 weeks training period. We measure the inclusion rate-i.e. the proportion of participants invited to participate who enroll into the study-and distinguish between those who refuse, did not respond or who were willing but excluded (volunteered but did not meet the study inclusion criteria). For attrition, we measure the number of participants lost at follow-up. For adherence to the intervention, we record engagement with the intervention, e.g. compliance with all trainings. There are 18 Virtual Reality video game training sessions possible for each individual.

SECONDARY OUTCOMES:
Cortico-muscular coherence (CMC); neuronal communication between Motor cortical areas and muscles | Immediately post-intervention following six weeks of intervention.
  CMC is essentially a measure giving an output value ranging from 0 to 1, the higher the number the better is the neuronal communication between motor cortical areas and muscles. Additionally, we will calculate when the coherence estimates will be significantly larger than zero at a specific labda exceeding a confidence limit (CL) with probability of 95% (α=0.05), with the following equation (2), where alpha denotes the significance Level.
gait kinematics; spatio-temporal Parameters of gait | Immediately post-intervention following six weeks of intervention.
  gait kinematics measured with the Physilog® (Gait up Sàrl, Lausanne, Switzerland) via wearable movement sensors (50×37×9.2mm, 19gramms, anatomical curved shape) containing inertial sensors.
Tegner Activity Score (TAS) | Immediately post-intervention following six weeks of intervention.
  Graduated list of activities of daily living, recreation, and competitive sports. Patient selects the level of participation that best describes their current level of activity. A score of 10 is assigned based on the level of activity that the patient selects. Score 0 represents "sick leave or disability pension because of knee problems," a score of 10 corresponds to participation in national and international elite competitive sports. Has been used more recently as a patient-completed questionnaire. A score of 10 is assigned based on the level of activity that the patient selects as best representing their current activity level. Possible score range: 0-10. Higher scores represent participation in higher-level activities.
International Knee Documentation Committee (IKDC) outcome | Immediately post-intervention following six weeks of intervention.
  a knee-specific patient-reported outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Hönggerberg, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Only anonymised data will be shared